CLINICAL TRIAL: NCT00888992
Title: Technology-Enhanced Quitline Services to Prevent Smoking Relapse
Acronym: TEQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Consumer Wellness Solutions (Industry); Kaiser Foundation Hospitals, Center for Health Research (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0812-77B; 1R01CA138936-01 (NIH)
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Smoking Cessation
Keywords: Smoking; Cessation; Quitline; Counseling
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (No Intervention): Receive the usual care provided in Alere Wellbeing's Quit For Life® program. The program includes 5 telephone counseling calls.
- Group B (Experimental)
  Interventions: Behavioral: Quitline Service + 10 automated monitoring calls
- Group C (Experimental)
  Interventions: Behavioral: Quitline service + 20 automated monitoring calls

INTERVENTIONS:
Behavioral: Quitline Service + 10 automated monitoring calls — This group will receive the usual care provided in Alere Wellbeing's Quit For Life® program. The program includes 5 telephone counseling calls. In addition, participants receive 10 automated telephone monitoring calls to help them stay off cigarettes. The automated call schedule will be two calls per a week for 2 weeks, then once a week for 6 weeks. Participants whose answers indicate that they may be having trouble quitting smoking will be automatically connected to a Quit Coach for individualized relapse prevention counseling.
  Arms: Group B
Behavioral: Quitline service + 20 automated monitoring calls — This group will receive the usual care provided in Alere Wellbeing's Quit For Life® program. The program includes 5 telephone counseling calls. In addition, participants receive 20 automated telephone monitoring calls to help them stay off cigarettes. The automated call schedule will be one automated call a day for 2 weeks, then once a week for 6 weeks. Participants whose answers indicate that they may be having trouble quitting smoking will be automatically connected to a Quit Coach for individualized relapse prevention counseling.
  Arms: Group C

SUMMARY:
The purpose of this study is to see if automated telephone monitoring will enhance existing quitline services, such as Alere Wellbeing's Quit For Life program, and help people quit smoking. If successful, this intervention could be incorporated into existing quitline protocols and delivered to millions of people who are trying to quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Enrolled in Free & Clear, Inc. services
* Self-reported abstinence for at least 24 hours at the quit date call
* Able to read and speak English
* Personal access to a touch-tone telephone or cellular telephone

Exclusion Criteria:

* Have not stopped smoking for 24 hours
* Currently incarcerated
* Currently participating in any other smoking cessation research
* Live in same household as another study participant
* Participated in the Alere Wellbeing Quit for Life Program within the last 6 months
* Were previously enrolled in this study even if they repeat the smoking cessation program during the accrual period
* Hearing impaired enrollees receiving Free & Clear services via telecommunications devices for the deaf (TDD) will be excluded from the study as the IVR technology currently does not have this capability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1785 (Actual)
Dates: Start 2010-04; Primary Completion 2013-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Participant smoking status. | 6 and 12 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Anna M McDaniel, PhD RN FAAN, Principal Investigator — Indiana University; Susan Zbikowski, PhD, Principal Investigator — Consumer Wellness Solutions; Katie Witkiewitz, PhD, Principal Investigator — University of New Mexico; Jeffery Fellows, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Alere Wellbeing (formally known as Free & Clear, Inc.), Seattle, Washington, United States

REFERENCES:
- [Derived] McDaniel AM, Vickerman KA, Stump TE, Monahan PO, Fellows JL, Weaver MT, Carlini BH, Champion VL, Zbikowski SM. A randomised controlled trial to prevent smoking relapse among recently quit smokers enrolled in employer and health plan sponsored quitlines. BMJ Open. 2015 Jun 29;5(6):e007260. doi: 10.1136/bmjopen-2014-007260. PMID 26124508